CLINICAL TRIAL: NCT03050918
Title: A Pragmatic, Randomized, Controlled Trial Examining the Effectiveness of a Hospital Discharge Follow-up Phone Call Program
Brief Title: Discharge Follow-up Phone Call Program
Acronym: FUTR-30
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Maame Yaa A. B. Yiadom, MD, MPH, MSCI, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 170019
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Results first posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Discharge Follow-up Phone Calls

STUDY DESIGN:
Intervention Model Description: This is a single center, pragmatic, randomized, controlled clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phone Call Group (Intervention Arm) (Active Comparator): Follow-up phone call intervention: Patients will receive the first call attempt within 72 hours of hospital discharge with a maximum of 3 call attempts by the study nurse made up until post-discharge day 7. The semi-structured script embedded within the program specific electronic health record Discharge Phone Call Starform is used to guide a conversation to obtain information on potential causes of hospital readmission that can be identified and addressed to improve each patient's transition to outpatient care.
  Interventions: Behavioral: Follow-up Phone Call
- Usual Care Group (Control Arm) (No Intervention): Patients assigned to the control group receive standard discharge planning and follow-up per the usual care of their medical providers.

INTERVENTIONS:
Behavioral: Follow-up Phone Call — Patients will receive a first call attempt within 72 hours discharge.
  Arms: Phone Call Group (Intervention Arm)

SUMMARY:
The goal of this project is to quantify the impact of post-hospital discharge follow-up phone calls on hospital readmission, ED visits, patient satisfaction, and mortality in a general medicine inpatient population. We will obtain exploratory information on patient sub-groups at high risk for hospital readmission and on those experiencing high benefit from the follow-up phone call intervention. In addition, we will obtain data on discharge plan implementation assistance needed to support a successful transition from inpatient to outpatient care among those reached by the intervention phone call.

DETAILED DESCRIPTION:
RATIONALE

In the current medical literature, it is unclear how follow-up calls influence these outcomes in a general medical population. Some studies have attempted to address this question, but are limited in that they target very specific patient populations, are of insufficient quality, or evaluated follow-up calls as part of a larger care bundle. We will conduct a high quality, real-time clinical care study to determine the efficacy of a follow-up phone call program.

STUDY DESIGN

This is a single center, pragmatic, randomized, controlled clinical trial to investigate whether a structured post-hospital discharge follow-up phone call can improve patients' transition from in-hospital to outpatient care and improve satisfaction with their care. We will also identify the discharge implementation assistance given to those in the intervention (Phone Call) group.

Outcome Measures Primary outcome for this study is readmission event rate within 30 days. Secondary outcomes include patient satisfaction which will be measured as mean Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) patient satisfaction scores, all cause VUMC emergency department (ED) visits, the need for assistance with discharge plan implementation, and 30 day mortality.

ELIGIBILITY:
Inclusion Criteria:

* VUMC patients discharged after an inpatient status hospital stay on a general medicine service.

Exclusion Criteria:

* patients who experience in-hospital death
* patient discharged to any post-acute care facility or inpatient hospice
* left the hospital against medical advice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3054 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2018-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maame Yaa Yiadom, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, semi-structured intervention script, randomization code, data flow design have been published to share with other investigators.
  Individual study data will be available to other investigators upon request per details below.
Supporting Information: Study Protocol
Time Frame: The study protocol was published in BMJ Open in 2017 (Yiadom MYAB, Domenico H, Byrne D, et al Randomised controlled pragmatic clinical trial evaluating the effectiveness of a discharge follow-up phone call on 30-day hospital readmissions: balancing pragmatic and explanatory design considerations BMJ Open 2018;8:e019600. doi: 10.1136/bmjopen-2017-019600)
  A full de-identified version of the database including participate data for this study will be available to other investigators upon request after consideration of their proposed use for the data. We are happy to begin accepting requests starting 12 months following the publication of the manuscript including study results.
Access Criteria: All requests should be directed to the corresponding author (maya.yiadom@vumc.org).

REFERENCES:
- [Derived] Yiadom MYAB, Domenico HJ, Byrne DW, Hasselblad M, Kripalani S, Choma N, Tucker-Marlow S, Gatto CL, Wang L, Bhatia MC, Morrison J, Harrell FE, Hartert TV, Lindsell CJ, Bernard GR. Impact of a Follow-up Telephone Call Program on 30-Day Readmissions (FUTR-30): A Pragmatic Randomized Controlled Real-world Effectiveness Trial. Med Care. 2020 Sep;58(9):785-792. doi: 10.1097/MLR.0000000000001353. PMID 32732787
- [Derived] Yiadom MYAB, Domenico H, Byrne D, Hasselblad MM, Gatto CL, Kripalani S, Choma N, Tucker S, Wang L, Bhatia MC, Morrison J, Harrell FE, Hartert T, Bernard G. Randomised controlled pragmatic clinical trial evaluating the effectiveness of a discharge follow-up phone call on 30-day hospital readmissions: balancing pragmatic and explanatory design considerations. BMJ Open. 2018 Feb 14;8(2):e019600. doi: 10.1136/bmjopen-2017-019600. PMID 29444787

RESULTS

PARTICIPANT FLOW:
Groups:
- Phone Call Group (Intervention Arm): Follow-up phone call program: Patients will receive the first call attempt within 72 hours of hospital discharge with a maximum of 3 call attempts by the study nurse made up until post-discharge day 7. The semi-structured script embedded within the program specific electronic health record Discharge Phone Call Starform is used to guide a conversation to obtain information on potential causes of hospital readmission that can be identified and addressed to improve each patient's transition to outpatient care.
Period: Overall Study
Arm/Group | Phone Call Group (Intervention Arm) | Usual Care Group (Control Arm)
Started | 1534 | 1520
Completed | 1534 | 1520
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phone Call Group (Intervention Arm) | Usual Care Group (Control Arm) | Total
Number analyzed (Participants) | 1534 | 1520 | 3054
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (17.7) | 53.4 (18.1) | 52.9 (17.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 761 | 749 | 1510
  Male | 773 | 771 | 1544
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 323 | 314 | 637
  White | 1164 | 1158 | 2322
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 47 | 48 | 95
Region of Enrollment [Number; unit: participants]
  United States | 1534 | 1520 | 3054
Highest Education/grade completed [Mean (Standard Deviation); unit: grade level in years] | 13.2 (3.5) | 12.9 (3.5) | 13.07 (3.54)
Brief Health Literacy Score [Mean (Standard Deviation); unit: scores on a scale] — Measures health literacy and patients ability to act as an independent agent for their own medical care. A score of <10 is considered to be inadequate to act alone as an independent agent for their own medical care and can identify patients that need assistance. Total score can range from 3 (low health literacy) to 15 (high health literacy).
  scores on a scale | 11.8 (3.5) | 12.0 (3.5) | 11.91 (3.47)
Established Primary Care Provider [Count of Participants; unit: Participants] | 982 | 1018 | 2000
Hospital Length of Stay [Mean (Standard Deviation); unit: days] | 4.5 (4.3) | 4.6 (4.7) | 4.54 (4.48)
Any time on Intensive Care Unit during stay [Count of Participants; unit: Participants] | 281 | 308 | 589
Predicted Re-admission risk before discharge [Mean (Standard Deviation); unit: percent risk] — The Predicted Readmission Risk Before Discharge is the result of a real-time predictive model embedded and displayed in the Vanderbilt Adult Hospital's electronic health record (EHR). It was developed through a collaboration between the Medical Center's Office of Quality Safety and Risk Prevention and the Vanderbilt Institute for Clinical and Translational Research and embedded into the EHR. The range for the predicted readmission risk is 0-100 (percent). Higher numbers indicate higher risk of re-admission.
  percent risk | 24.4 (15.9) | 23.4 (14.2) | 23.9 (15.1)
In-patient Admission in prior 6 months [Count of Participants; unit: Participants] | 483 | 461 | 944
Mean number of In-Patient admissions in the prior 6 months [Mean (Standard Deviation); unit: in-patient admissions] | 0.6 (1.2) | 0.6 (1.1) | 0.6 (1.184)
CMS Re-admission Penalty Group: COPD Exacerbation [Count of Participants; unit: Participants] | 320 | 327 | 647
CMS Re-admission Penalty Group: Pneumonia [Count of Participants; unit: Participants] | 384 | 371 | 755
CMS Re-admission Penalty Group: Heart Failure [Count of Participants; unit: Participants] | 234 | 234 | 468
CMS Re-admission Penalty Group: Acute Myocardial Infarction [Count of Participants; unit: Participants] | 79 | 80 | 159
CMS Re-admission Penalty Group: Stroke [Count of Participants; unit: Participants] | 22 | 37 | 59
CMS Re-admission Penalty Group: Total hip/knee [Count of Participants; unit: Participants] — Re-admission for Elective Primary Total Hip Arthroplasty and/or Total Knee Arthroplasty (THA/TKA)
  Participants | 1 | 1 | 2
CMS Re-admission Penalty Group: Coronary Artery Bypass Graph [Count of Participants; unit: Participants] | 0 | 0 | 0
CMS Re-admission Penalty Group: None [Count of Participants; unit: Participants] | 836 | 825 | 1661

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With In-patient Re-admissions
Description: Number of participants with in-patient re-admissions
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phone Call Group (Intervention Arm) | Usual Care Group (Control Arm)
Number analyzed (Participants) | 1534 | 1520
Participants | 228 | 232
Statistical Analysis 1: Comparison: Phone Call Group (Intervention Arm) vs Usual Care Group (Control Arm); Test type: Superiority; p = .05, Wilcoxon (Mann-Whitney) — we used the O'Brian-Fleming α-spending function, allowing for an α-level of significance of 0.005 and 0.048 for the interim and final analyses, respectively

2. Secondary Outcome: Patient Satisfaction: Experience
Description: Measured as mean Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) patient satisfaction scores. Higher scores indicate more patient satisfaction. Range is 0-9 with 9 being the most satisfied.
Time Frame: Within 60 days of Discharge
Population: Patient experience data were retrieved from the hospital quality and patient safety office at 60 days, but assessment was administered via a survey sent to patients at their home after hospital discharge. Scores are based on the number of surveys returned
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phone Call Group (Intervention Arm) | Usual Care Group (Control Arm)
Number analyzed (Participants) | 227 | 249
score on a scale | 8.2 (1.8) | 8.3 (1.4)
Statistical Analysis 1: Comparison: Phone Call Group (Intervention Arm) vs Usual Care Group (Control Arm); Test type: Superiority; p = 0.05, Chi-squared — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Phone Call Group (Intervention Arm) vs Usual Care Group (Control Arm); Test type: Superiority; p = .05, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Patient Satisfaction: Likelihood to Recommend the Facility (Top Box Rating)
Description: Measured as mean Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) patient satisfaction scores. Number of patients that reported a score of 3. Range is 0-3 with 3 being highest satisfaction.
Time Frame: Within 60 days of Discharge
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phone Call Group (Intervention Arm) | Usual Care Group (Control Arm)
Number analyzed (Participants) | 227 | 247
Participants | 168 | 193
Statistical Analysis 1: Comparison: Phone Call Group (Intervention Arm) vs Usual Care Group (Control Arm); Test type: Superiority; p = 0.05, Chi-squared — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Phone Call Group (Intervention Arm) vs Usual Care Group (Control Arm); Test type: Superiority; p = .05, Chi-squared — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Patient Satisfaction: Hospital Experience (Top Box Rating)
Description: Measured as mean Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) patient satisfaction scores. Number of patients that rated the Hospital Experience as 9. Scale range is 0-9. Higher scores indicate more patient satisfaction.
Time Frame: Within 60 days of Discharge
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phone Call Group (Intervention Arm) | Usual Care Group (Control Arm)
Number analyzed (Participants) | 227 | 249
Participants | 155 | 173
Statistical Analysis 1: Comparison: Phone Call Group (Intervention Arm) vs Usual Care Group (Control Arm); Test type: Superiority; p = .05, Chi-squared — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Patient Satisfaction: Likelihood to Recommend the Facility
Description: Measured as mean Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) patient satisfaction scores. Scale range is 0-3. Higher scores indicate more patient satisfaction.
Time Frame: Within 60 days of Discharge
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phone Call Group (Intervention Arm) | Usual Care Group (Control Arm)
Number analyzed (Participants) | 227 | 247
score on a scale | 2.7 (.7) | 2.7 (.6)
Statistical Analysis 1: Comparison: Phone Call Group (Intervention Arm) vs Usual Care Group (Control Arm); Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: VUMC Emergency Department (ED) Visits
Description: All cause ED visits following discharge
Time Frame: 30 days
Measure: Number; unit: ED visits
Arm/Group | Phone Call Group (Intervention Arm) | Usual Care Group (Control Arm)
Number analyzed (Participants) | 1534 | 1520
ED visits | 93 | 82
Statistical Analysis 1: Comparison: Phone Call Group (Intervention Arm) vs Usual Care Group (Control Arm); Test type: Superiority; p = 0.05, Chi-squared — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Patient Received Discharge Plan Implementation Assistance
Description: Need for assistance in implementing discharge plan
Time Frame: 30 days
Population: Discharge plan implementation assistance was offered as part of the intervention and not to the control group.
Measure: Count of Participants; unit: Participants
Arm/Group | Phone Call Group (Intervention Arm) | Usual Care Group (Control Arm)
Number analyzed (Participants) | 1534 | 0
Participants | 463 | 0

8. Secondary Outcome: Mortality
Description: All cause mortality
Time Frame: 30 days
Population: Thirty-day mortality data was retrieved from the EHR data repository after a 120-day lag to capture delayed reporting.
Measure: Count of Participants; unit: Participants
Arm/Group | Phone Call Group (Intervention Arm) | Usual Care Group (Control Arm)
Number analyzed (Participants) | 1534 | 1520
Participants | 68 | 75
Statistical Analysis 1: Comparison: Phone Call Group (Intervention Arm) vs Usual Care Group (Control Arm); Test type: Superiority; p = 0.05, Chi-squared — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse Events were evaluated in 3 ways: 1) all-cause mortality, 2) reviewing a 10% sample of the Phone Call Nurse's daily reports, and 3) reviewing the Phone Call Program office's internal quality assessment for evidence the intervention may introduce harm.
Arm/Group | Phone Call Group (Intervention Arm) | Usual Care Group (Control Arm)
All-Cause Mortality (participants affected / at risk) | 68/1534 | 75/1520
Serious Adverse Events (participants affected / at risk) | 0/1534 | 0/1520
Other Adverse Events (participants affected / at risk) | 0/1534 | 0/1520

LIMITATIONS AND CAVEATS:
A data lag due to limited national electronic health record informatics connectivity prevents us from tracking adverse events documented outside of our facility. Unmeasured outcomes should be equally distributed between the randomized groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT03050918/Prot_SAP_000.pdf